CLINICAL TRIAL: NCT05951855
Title: Selinexor in Combination With Chidamide in Unfit Relapsed/Refractory Acute Leukemia: a Phase 2, Single-Arm, Open-Label, Multi-Center Prospective Study.
Brief Title: Study of Selinexor Combined With Chidamide in Relapsed/Refractory Acute Leukemia (AML) Patients
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Soochow University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Selinexor+ Chidamide
Record Dates: First submitted 2023-06-24; First posted 2023-07-19 (Actual); Last update posted 2023-07-19 (Actual); Status verified 2022-08

CONDITIONS: Acute Myeloid Leukemia (Relapsed/Refractory)
Keywords: relapsed/refractory; AML; selinexor and chidamide
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Recurrence | interventions — selinexor; N-(2-amino-5-fluorobenzyl)-4-(N-(pyridine-3-acrylyl)aminomethyl)benzamide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Selinexor combined with chidamide (Experimental): R/R AML who are ineligible for intensive chemotherapy will receive selinexor in combination with chidamide, 28 days per cycle, Selinexor will be used as 40 or 60mg BIW for two weeks, and chidamide will be used as 10mg/d from day 1 to 28. Depending on the level of recovery, patients will either be forced to come off study or have the option to continue the medication, receive maintenance therapy, or pursue an allogeneic stem cell transplant.
  Interventions: Drug: Selinexor; Drug: Chidamide

INTERVENTIONS:
Drug: Selinexor — Selinexor 60mg/day, weight≥70kg (40mg/day, weight<70kg) orally on d1,4,8,11,
  Other Names: X
Drug: Chidamide — Chidamide 10mg/day, orally on day 1 to 28
  Other Names: C

SUMMARY:
This is a prospective, single-arm, multi-center clinical trial to evaluate the efficacy and safety of selinexor combined with chidamide in the treatment of unfit R/R AML.

DETAILED DESCRIPTION:
This protocol corresponds to a multicenter, open-label, single arm, prospective study designed to determine the efficacy and safety of selinexor in combination with chidamide for unfit R/R AML.

Selinexor will be given orally at 40 or 60mg on d1,4,8,11; Chidamide will be given orally at 10mg on d1-28; 28 days per cycle. patients can receive transplants at any time once they achieved complete remission and other patients will continue to receive treatment until disease progression or unacceptable toxic effects. After completion of study treatment, participants are followed up every 3 to 6 months for up to 2 years.

Study design allows 42 patients.

ELIGIBILITY:
Inclusion Criteria:

1. Men and women aged 18 to 75 years old.
2. Diagnosis of relapsed or refractory AML (defined according to the the World Health Organization [WHO] 2016 criteria) of any type except for acute promyelocytic leukemia (APL; AML M3).
3. Eastern Cooperative Oncology Group (ECOG) performance status of 2-3.
4. Patients whose expecting survival time will be more than 3 months.
5. One of the serious heart, lung, liver, kidney disease:

   1. Cardiac history of Congestive Heart Failure (CHF) requiring treatment or Ejection Fraction <= 50% or chronic stable angina;
   2. Diffusing capacity of the Lung for Carbon Monoxide (DLCO) <= 65% or Forced Expiratory Volume in 1 second (FEV1) <= 65%;
   3. Moderate hepatic impairment with total bilirubin > 1.5 to <= 3.0 × Upper Limit of Normal (ULN);
   4. Creatinine clearance >= 30 mL/min to < 45 ml/min;
6. Other comorbidities that the physician judges to be incompatible with intensive chemotherapy.
7. Patients who had not received radiotherapy, chemotherapy, targeted therapy within one week before enrollment.
8. Fertile women and men whose partner is of childbearing potential or pregnant should agree to practice complete abstinence or to use a condom during therapy and dose interruptions and for 90 days after the last treatment.
9. Patients who are suitable for intensive chemotherapy but refuse it.
10. Patients who have known and voluntarily signed the informed consent (ICF).

Exclusion Criteria:

1. History of any malignancies prior to study entry with exception noted in the protocol.
2. Patients who had previously been treated with selinexor and/or chidamide.
3. Patients with APL/AML M3, or t(9;22)(q34.1;q11.2); BCR-ABL1 positive AML.
4. Absolute white blood cell count >=100*10^9/L.
5. Persistent toxicity due to previous chemotherapy or radiotherapy did not recover to 2 grade.
6. Presence of CNS leukemia.
7. Patients who had undergone cardiac angioplasty or stent implantation within 12 months before signing the informed consent form, or had myocardial infarction or instability history of defined angina or other clinically significant cardiac events.
8. Ucontrolled active infection (including bacterial, fungal or viral infections) and bleeding from internal organs.
9. Pregnant and lactating women.
10. Participated in any other clinical trials within 3 months before signing the informed consent form.
11. Patients who are unsuitable for this study judged by clinicians.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2023-03-01 (Actual); Primary Completion 2024-09-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Number of Participants With ORR | 28 days after study treatment
  Defined as complete response (CR) + CR with incomplete blood count recovery (CRi) + morphologic leukemia-free state (MLFS) + partial response (PR).

SECONDARY OUTCOMES:
Duration of Response (DOR) | 2 years
  Defined as time, in months, from initial response (CR+CRi+PR+MLFS) until the date of a disease progression
Event-free survival (EFS) | Time from registration to event, max 3 years
  Defined as the number of days from the date of treatment initiation (i.e., course 1 day 1) to the date of documented treatment failure, relapses from CR, or death from any cause, whichever occurs first. Will be calculated for all patients. Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.
Overall Survival (OS) | Time from registration to event, max 3 years
  Calculated from the date of informed consent to the date of death. Patients still alive at the end of follow-up were censored at the last date of follow-up. Estimated using Kaplan-Meier method. Log-rank tests will be used to compare among subgroups of patients.
Number of Adverse Events (AE) | continuously from first administration of study drug untill 30 days after last study treatment. (approximately up to 1 year)
  Adverse events are evaluated with CTCAE V5.0.

CONTACTS AND LOCATIONS:
Overall Officials: Huiying Qiu, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University
Locations (1):
- The First Affiliated Hospital of Soochow University, Suzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No